CLINICAL TRIAL: NCT06400004
Title: A Phase III Crossover Study to Evaluate Bolus Versus Continuous Infusion of Lumason® in Patients With Suboptimal Unenhanced Echocardiography
Brief Title: Lumason® Infusion vs. Bolus Administrations
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: BR1-149
Record Dates: First submitted 2024-04-23; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases | interventions — Suspensions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bolus administration (Active Comparator): Bolus administration of 2 mL undiluted Lumason®
  Interventions: Drug: Sulfur Hexafluoride Lipid Type A Microspheres 25 MG Injection Powder for Suspension [LUMASON]
- Continuous infusion (Experimental): Continuous infusion of 8 mL of diluted Lumason®
  Interventions: Drug: Lumason

INTERVENTIONS:
Drug: Sulfur Hexafluoride Lipid Type A Microspheres 25 MG Injection Powder for Suspension [LUMASON] — Bolus administration of 2 mL undiluted Lumason®, to be administered in 20 seconds
  Other Names: Bolus Administration
  Arms: Bolus administration
Drug: Lumason — Continuous infusion of 8 mL of diluted Lumason® (4 mL of Lumason® diluted in 4 mL of saline) at a rate of 1.0 mL/min
  Other Names: Infusion Administration
  Arms: Continuous infusion

SUMMARY:
A phase III study designed as a randomized, within-patient comparison of continuous infusion of diluted Lumason® versus the bolus administration of undiluted Lumason® for degree of LVO and assessment of LV EBD (co-primary endpoints).

DETAILED DESCRIPTION:
This is a phase III study designed as a randomized, within-patient comparison of continuous infusion of diluted Lumason® versus the bolus administration of undiluted Lumason® for degree of LVO and assessment of LV EBD (co-primary endpoints). The study will enroll patients with suboptimal LV EBD defined as ≥2 adjacent segments in any apical view that cannot be visualized at pre-contrast echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18-years old;
* Have suboptimal LV EBD, defined as ≥2 adjacent segments in any apical view that cannot be visualized, at pre-contrast echocardiogram;
* Provide their written informed consent and are willing to comply with protocol requirements.

Exclusion Criteria:

* Patient has severe congestive heart failure (class IV according to the classification of the New York Heart Association);
* Patient has uncontrolled angina (i.e., uncontrolled on medication);
* Patient had a recent myocardial infarction (within the last 3 days and not stabilized);
* Patient has severe arrhythmia, that in the opinion of the Investigator, would interfere with the study conduct;
* Patient has severe pulmonary hypertension, that in the opinion of the Investigator, would interfere with the study conduct;
* Patient had been treated with any other contrast medium, either intravascular or orally, within 48 hours prior to the first administration;
* Has any known allergy to one or more of the ingredients of the investigational product;
* Is pregnant or lactating. Exclude the possibility of pregnancy by: testing on site (serum or urine βHCG) prior to the start of investigational product administration; surgical history (e.g., tubal ligation or hysterectomy); post-menopausal with a minimum 1 year without menses;
* Has previously entered the study or have received any other investigational drug within 30 days prior to admission in this study;
* Is determined by the Investigator that the patient is clinically unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Adequate LV EBD Score | 2-3 Hours
  Compare the proportion of patients with adequate LV EBD score for infusion vs. bolus administrations in patients with suboptimal left ventricular endocardial border delineation at unenhanced echocardiography.
Adequate LV Opacification | 2-3 Hours
  Compare the proportion of patients with adequate LV opacification for infusion vs. bolus administrations in patients with suboptimal left ventricular endocardial border delineation at unenhanced echocardiography.

SECONDARY OUTCOMES:
Clinically useful LVO | 2-3 Hours
  To compare the duration of clinically useful LVO in infusion vs. bolus administrations in terms of duration
Adverse events | 24 Hours
  Compare adverse event rate after infusion vs. bolus administrations

CONTACTS AND LOCATIONS:
Overall Officials: Jose Banchs, MD, Study Director — Sr. Medical Director
Locations (3):
- United States (3):
  - Piedmont Heart Institute, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Oregon Health and Sciences University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No